CLINICAL TRIAL: NCT04666467
Title: Early Feasibility EXperience of Posterior Leaflet RestOration to REduce Functional Mitral Regurgitation (EXPLORE FMR)
Brief Title: Early Feasibility Study of the PLAR Implant and Delivery System to Treat Functional Mitral Regurgitation ( EXPLORE FMR )
Acronym: EXPLORE FMR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study device refinement
Sponsor: Polares Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 202002
Record Dates: First submitted 2020-12-01; First posted 2020-12-14 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Functional Mitral Regurgitation

STUDY DESIGN:
Intervention Model Description: Single arm registry
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single-arm study of PLAR Implant and Delivery System (Experimental): All enrolled patients will receive the study device
  Interventions: Device: Transcatheter mitral valve repair

INTERVENTIONS:
Device: Transcatheter mitral valve repair — Transvenous approach with a transeptal puncture to place the study device
  Other Names: TMVr

SUMMARY:
An early feasibility study to evaluate the safety and feasibility of the PLAR Implant and Delivery System to treat severe functional mitral regurgitation and to gather preliminary data on its performance thereby providing guidance for future clinical development. The study is a single-arm registry with the last follow-up visit at 5 years post-intervention. The study will enroll up to 10 patients at up to 4 centers in North America.

DETAILED DESCRIPTION:
Percutaneous approaches to treat MR promise to provide a sufficient reduction in MR without the risks typically associated with open heart surgery. Furthermore there is an unmet clinical need for patients with severe MR who are refused or denied surgery due to high risk. Percutaneous therapy provides a novel alternative treatment option for these patients with the aim of reducing morbidity and mortality over and above current medical therapy. The Polares Medical PLAR Implant and Delivery System is a catheter-based technology designed to permanently implant a prosthesis using a transvenous / transseptal approach to augment the posterior mitral valve leaflet and improve coaptation of the mitral valve. Approved edge-to-edge repair has already been shown to be a viable alternative for high risk MR patients. However treatment with these devices is limited to specific anatomies and often requires multiple devices which increases clinical risk, adds to procedural time, and can result in residual MR. The PLAR Implant and Delivery System has been designed to overcome and mitigate some of these shortfalls.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Greater than moderate functional mitral regurgitation (Grade 3+ or higher) as confirmed by transesophageal echocardiography (TEE) within 90 days prior to study procedure
3. Patient must present with an STS Score less than 10%
4. High surgical risk for conventional mitral repair or replacement due to morphological criteria (e.g. leaflet or annulus calcifications), but operable, as assessed by the local heart team comprised of a cardiac surgeon experienced in mitral valve surgery and a cardiologist experienced in treating mitral valve disease and heart failure
5. Patient is approved by an independent Patient Eligibility Committee
6. New York Heart Association (NYHA) Functional Class III or IV
7. Patient willing to participate in study and sign the IRB/EC-approved informed consent
8. Treating physician and patient agree that patient is able to return for all required post-procedure follow-up visits
9. Women of child-bearing potential have a negative pregnancy test

Exclusion Criteria:

1. Severe tricuspid regurgitation
2. Severe aortic stenosis or insufficiency
3. Severe mitral annulus calcification
4. Diseased mitral anterior leaflet such as flail / prolapse/ heavy calcification
5. Implanted vena cava filter
6. Femoral veins with severe angulation and calcification
7. Contraindication for transesophageal echocardiography (TEE) or MDCT scan
8. Active infection or endocarditis
9. Previous mitral valve surgery
10. Prior orthotopic heart transplantation
11. Pulmonary artery systolic hypertension > 70mmHg
12. Evidence of intra-cardiac, inferior vena cava (IVC) or femoral venous thrombus
13. Left ventricular ejection fraction (LVEF) < 30%
14. Implant or revision of any pacing device < 30 days prior to intervention
15. Symptomatic coronary artery disease treated < 30 days prior to study procedure
16. Myocardial infarction requiring intervention < 30 days prior to study procedure
17. Infiltrative cardiomyopathies (e.g., amyloidosis, hemochromatosis, sarcoidosis), hypertrophic or restrictive cardiomyopathies, and constrictive pericarditis
18. Active peptic ulcer or upper gastrointestinal bleeding < 90 days prior to study procedure
19. Stroke < 180 days prior to study procedure
20. Severe renal insufficiency (creatinine > 3.0 mg/dL) or patient requiring dialysis
21. Cardiogenic shock at time of enrollment
22. Hemodynamic instability requiring inotropic support or mechanical heart assistance
23. Concurrent medical condition with a life expectancy of less than 2 years
24. Pregnancy at time of enrollment
25. History of bleeding diathesis or coagulopathy or leukopenia (WBC < 3,000 mcL) or acute anemia (Hb < 9 g/dL) or thrombocytopenia (platelets < 50,000 cells mcL)
26. Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine or clopidogrel, nitinol, tantalum or allergy to contrast agents that cannot be pre-medicated
27. Emergency situations
28. Severe dementia or lack of capacity due to conditions that result in either inability to provide informed consent for the trial/procedure, prevent independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up assessments
29. Company employees or their immediate family members
30. Patient is under guardianship
31. Patient is participating in another clinical study for which follow-up is currently ongoing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of all-cause mortality | 30-days
  Primary safety outcome
Incidence of change from baseline to moderate or less mitral regurgitation (Grade 2+ or less) as evaluated by 2D TTE | 30-days
  Primary performance endpoint

SECONDARY OUTCOMES:
Rate of major safety events as defined by MVARC2 definitions | 30 days, at 6 and 12 months, and at 2 - 5 years
  Secondary safety endpoint
Technical success rate per MVARC2 definitions | Technical success is measured at exit from OR
  Absence of procedure mortality
  * Successful access, delivery and retrieval of investigation delivery system
  * Successful deployment and correct positioning of intended implant(s)
  * Freedom from emergency surgery/re-intervention related to device or access procedure
Procedure success rate per MVARC2 definitions | Procedure success is measured at 30 days post-intervention
  Device success and absence of major device or procedure-related serious adverse events as below:
  * Death
  * Stroke
  * Life-threatening bleed
  * Major vascular complication
  * Major cardiac structural complication
  * Stage 2 or 3 AKI
  * MI or coronary ischemia requiring PCI or CABG
  * Shock, heart or respiratory failure requiring IV vasopressors, mechanical intervention or prolonged intubation
  * Valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention
Device success rate per MVARC 2 definitions (all must be present for success) | Device success is measured at 30 days, at 6 and 12 months, and at 2 - 5 years post-intervention
  * Absence of procedure mortality or stroke
  * Proper placement and positioning of device
  * Freedom from unplanned re-intervention related to device or access procedure
  * Continued intended safety and performance of the device:
    * No evidence of structural or functional failure
    * No device technical failure issues/complications
    * MR reduction to moderate or less without stenosis
Patient success rate per MVARC2 definitions (all must be present for success) | Patient success is measured at 12 months post-intervention
  * Device success
  * Patient returned to pre-procedure setting
  * No rehospitalization or reintervention for mitral regurgitation or heart failure
  * Functional improvement from baseline by one or more NYHA class
  * 6MWT improvement from baseline by 50 metres or more

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Brenton, Study Director — Polares Medical
Locations (1):
- Emory Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Clinical trial results will be shared with investigators once study is enrolled and trial data is prepared for presentation at a medical conference or for publication in a medical journal.